CLINICAL TRIAL: NCT01681992
Title: Immunogenicity and Safety Study of GSK Biologicals' Priorix Vaccine (209762) at an End of Shelf-life Potency Compared to Merck & Co., Inc.'s Measles-mumps-rubella (MMR) Vaccine When Both Are Given on a 2-dose Schedule to Healthy Children in Their 2nd Year of Life
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Combined Measles-mumps-rubella (MMR) Vaccine in Children in Their Second Year of Life
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 115649; 2011-004905-26 (EudraCT Number)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Measles; Mumps; Rubella; Measles-Mumps-Rubella Vaccine
Keywords: Safety; Measles, mumps and rubella diseases; Immunogenicity
MeSH Terms: conditions — Measles; Mumps; Rubella | interventions — Measles-Mumps-Rubella Vaccine; Rubella Vaccine; Chickenpox Vaccine; Hepatitis A Vaccines; 13-valent pneumococcal vaccine; CRM197 (non-toxic variant of diphtheria toxin)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (3):
- Inv_MMR_Min Group (Experimental): Subjects receive one dose of GlaxoSmithKline (GSK) Biologicals' measles, mumps, rubella (MMR) vaccine, Priorix (Inv_MMR), from a minimum potency lot (Inv_MMR_Min), co-administered with Varivax (VV) and Havrix (HAV) vaccines at Day 0. All US subjects are also co-administered Prevnar 13 (PCV-13) vaccine. Approximately 6 weeks later, at Day 42, subjects are administered a dose from a separate lot of the Inv_MMR vaccine (Inv_MMR_Release), for the second dose. Inv_MMR and VV vaccines are administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines are administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
  Interventions: Biological: Priorix; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13
- Inv_MMR_Med Group (Experimental): Subjects receive one dose of GlaxoSmithKline (GSK) Biologicals' measles, mumps, rubella (MMR) vaccine, Priorix (Inv_MMR), from a mid-range or medium potency lot (Inv_MMR_Med), co-administered with Varivax (VV) and Havrix (HAV) vaccines at Day 0. All US subjects are also co-administered Prevnar 13 (PCV-13) vaccine. Approximately 6 weeks later, at Day 42, subjects are administered a dose from a separate lot of the Inv_MMR vaccine (Inv_MMR_Release), for the second dose. Inv_MMR and VV vaccines are administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines are administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
  Interventions: Biological: Priorix; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13
- Com_MMR Group (Active Comparator): Subjects receive one dose of M-M-R II (Com_MMR) vaccine (Lot 1 or Lot 2), co-administered with Varivax (VV) and Havrix (HAV) vaccines at Day 0. All US subjects are also co-administered Prevnar 13 (PCV-13) vaccine. Approximately 6 weeks later, at Day 42, subjects are administered a dose of Com_MMR vaccine (Lot 1 or Lot 2), for the second dose. Com_MMR and VV vaccines are administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines are administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
  Interventions: Biological: M-M-R II; Biological: Varivax; Biological: Havrix; Biological: Prevnar 13

INTERVENTIONS:
Biological: Priorix — Subjects receive one dose of either minimum (Inv_MMR_Min) or medium (Inv_MMR_Med) potency lot at Day 0 and a dose of separate potency lot (Inv_MMR_Release) at Day 42, administered subcutaneously in the triceps region of the left arm.
  Other Names: GSK Biologicals' live attenuated measles; mumps; rubella vaccine
  Arms: Inv_MMR_Med Group; Inv_MMR_Min Group
Biological: M-M-R II — Subjects receive two doses of either Lot 1 or Lot 2, one at Day 0 and one at Day 42, administered subcutaneously in the triceps region of the left arm.
  Other Names: Merck & Co.; Inc.'s measles; mumps; rubella virus vaccine; live
  Arms: Com_MMR Group
Biological: Varivax — Subjects receive one dose co-administered subcutaneously with the study vaccines (Priorix and M-M-R II), in the triceps region of right arm, at Day 0.
  Other Names: Merck & Co.; Inc.'s varicella virus vaccine; live
Biological: Havrix — Subjects receive one dose co-administered intramuscularly with the study vaccines (Priorix and M-M-R II), in the anterolateral region of the right thigh, at Day 0.
  Other Names: GSK Biologicals' hepatitis A vaccine; inactivated
Biological: Prevnar 13 — US Subjects receive one dose co-administered intramuscularly with the study vaccines (Priorix and M-M-R II), in the anterolateral region of the left thigh, at Day 0.
  Other Names: Pfizer Inc.'s pneumococcal 13-valent conjugate vaccine (diphtheria CRM197 protein)

SUMMARY:
The purpose of this study is to evaluate end of shelf-life potency in terms of the immunogenicity and safety of GSK Biologicals' trivalent MMR vaccine, by comparing it to Merck & Co., Inc.'s MMR vaccine, which is approved for use in the United States (US).

DETAILED DESCRIPTION:
This trial is a Phase IIIA, randomized, observer-blind, controlled, multi-center, multi-country study with four parallel groups. This study will evaluate the immunogenicity and safety of GSK Biologicals' trivalent investigational MMR vaccine (referred to as Inv_MMR vaccine, throughout this document) in contrast to the US standard of care comparator vaccine (M-M-R II, Merck and Co., Inc., referred to as Com_MMR throughout this document) in children during their second year of life. The first dose of this two-dose study is designed to establish the end of shelf-life potency of Inv_MMR vaccine. The Inv_MMR vaccine will be given as one of two lots; one of a minimum potency, designated Inv_MMR_Min; and the other at a mid-range or medium potency designated Inv_MMR_Med to two groups. The second dose for both of these Inv_MMR groups will have a potency within the release range of the marketed vaccine. The Com_MMR vaccine will consist of two lots designated Com_MMR_L1 and Com_MMR_L2 and will be analyzed as pooled lots within the study. The first MMR vaccine dose will be co-administered with Varivax, Havrix and (in the US sub-cohort only) Prevnar 13 which are routinely administered to children of this age in the US.

ELIGIBILITY:
Inclusion Criteria:

* Male or female child between 12 and 15 months of age at the time of vaccination.
* The investigator believes that the parent(s) or Legally Acceptable Representative(s) (LAR(s)) of the child, can, and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the child.
* Child is in stable health as determined by investigator's clinical examination and assessment of child's medical history.

For US children only:

• Child that previously received a 3-dose series of Prevnar 13 with last dose at least 60 days prior to study entry.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine(s) during the period starting 30 days before the day of study vaccination or planned use during the entire study period.
* Concurrently participating in another clinical study, in which the child has been or will be exposed to an investigational or a non-investigational product. Chronic administration of immunosuppressants, or other immune-modifying drugs during the period starting 180 days prior to the first vaccine dose or any planned administration of immunosuppressive and immune-modifying drugs during the entire study.

  * Inhaled and topical steroids are allowed.
* Planned administration / administration of a vaccine not foreseen by the study protocol during the period starting 30 days prior to study vaccination at Visit 1 and ending at Visit 2 (or ending at Visit 3 for the US post-dose 2 sub-cohort). Please Note:

  * Inactivated influenza (Flu) vaccine and Haemophilus influenzae type b conjugate vaccine (Hib) vaccines may be given at any time during the study, including the day of study vaccination (Flu and Hib vaccines must be administered at a different location than the study vaccine/s).
  * Any age appropriate vaccine may be given starting at Visit 2 (or starting at Visit 3 for the US post-dose 2 sub-cohort), and anytime thereafter.
* Administration of immunoglobulins and/or any blood products during the period starting 180 days prior to study vaccination at Visit 1 or planned administration from the date of vaccination through the immunogenicity evaluation at Visit 2, or at Visit 3 for the US post-dose 2 sub-cohort.
* History of measles, mumps, rubella, varicella/zoster and/or hepatitis A diseases.
* Known exposure to measles, mumps, rubella and/or varicella/zoster during the period starting 30 days prior to the first study vaccination.
* Previous vaccination against measles, mumps, rubella, hepatitis A and/or varicella virus.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including hypersensitivity to neomycin, latex or gelatin.
* Blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Fever is defined as temperature ≥38°C/100.4°F by any age appropriate route. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection without fever.
* Active untreated tuberculosis based on medical history.
* Any other condition which, in the opinion of the Investigator, prevents the child from participating in the study.

For US children only:

• A child that previously received a fourth dose of any pneumococcal conjugate vaccine.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4538 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2015-02-03 (Actual); Study Completion 2015-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (72):
- United States (36):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Muncie, Indiana
  - GSK Investigational Site, New Albany, Indiana
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Annapolis, Maryland
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Frederick, Maryland
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Clyde, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Youngstown, Ohio
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Johnstown, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Springville, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Midlothian, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Ellensburg, Washington
- Czechia (12):
  - GSK Investigational Site, Benešov
  - GSK Investigational Site, Chlumec nad Cidlinou
  - GSK Investigational Site, Děčín
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Kladno
  - GSK Investigational Site, Liberec
  - GSK Investigational Site, Lipník nad Bečvou
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Odolena Voda
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
- Finland (5):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- Malaysia (3):
  - GSK Investigational Site, Kuala Terengganu
  - GSK Investigational Site, Kuching
  - GSK Investigational Site, Sibu
- Puerto Rico (3):
  - GSK Investigational Site, Guayama
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan
- Spain (10):
  - GSK Investigational Site, Antequera/Málaga
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, L'Eliana, Valencia
  - GSK Investigational Site, Manlleu
  - GSK Investigational Site, Quart de Poblet, Valencia
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Vic
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Pathum Thani

REFERENCES:
- [Background] MMR-161 Study Group. Immunogenicity and safety of measles-mumps-rubella vaccine at two different potency levels administered to healthy children aged 12-15 months: A phase III, randomized, non-inferiority trial. Vaccine. 2018 Sep 11;36(38):5781-5788. doi: 10.1016/j.vaccine.2018.07.076. Epub 2018 Aug 10. PMID 30104117

RESULTS

PARTICIPANT FLOW:
Recruitment Details: US sub-cohort: Subjects recruited in US and received Inv_MMR_Min or Inv_MMR_Med or Com_MMR (Lot 1 or 2) co-administered with Varivax (VV), Havrix (HAV) and Prevnar 13 (PCV-13) at Day 0. Non-US sub-cohort: Subjects recruited outside US and received Inv_MMR_Min or Inv_MMR_Med or Com_MMR (Lot 1 or 2) co-administered with VV and HAV at Day 0.
Pre-assignment Details: 4538 subjects were registered in the study. 3 subjects were excluded because of invalid Informed Consent Forms and 19 subjects received a subject number but were not vaccinated. Therefore, the number of subjects started is 4516.
Groups:
- Inv_MMR_Min Group: Subjects received one dose of GlaxoSmithKline (GSK) Biologicals' measles, mumps, rubella (MMR) vaccine, Priorix (Inv_MMR), from a minimum potency lot (Inv_MMR_Min), co-administered with Varivax (VV) and Havrix (HAV) vaccines at Day 0. All US subjects were also co-administered Prevnar 13 (PCV-13) vaccine. Approximately 6 weeks later, at Day 42, subjects were administered a dose from a separate lot of the Inv_MMR vaccine (Inv_MMR_Release), for the second dose. Inv_MMR and VV vaccines were administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- Inv_MMR_Med Group: Subjects received one dose of GlaxoSmithKline (GSK) Biologicals' measles, mumps, rubella (MMR) vaccine, Priorix (Inv_MMR), from a mid-range or medium potency lot (Inv_MMR_Med), co-administered with Varivax (VV) and Havrix (HAV) vaccines at Day 0. All US subjects were also co-administered Prevnar 13 (PCV-13) vaccine. Approximately 6 weeks later, at Day 42, subjects were administered a dose from a separate lot of the Inv_MMR vaccine (Inv_MMR_Release), for the second dose. Inv_MMR and VV vaccines were administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- Com_MMR Group: Subjects received one dose of M-M-R II (Com_MMR) vaccine (Lot 1 or Lot 2), co-administered with Varivax (VV) and Havrix (HAV) vaccines at Day 0. All US subjects were also co-administered Prevnar 13 (PCV-13) vaccine. Approximately 6 weeks later, at Day 42, subjects were administered a dose of Com_MMR vaccine (Lot 1 or Lot 2), for the second dose. Com_MMR and VV vaccines were administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
Period: Overall Study
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Started | 1493 | 1497 | 1526
Completed | 1427 | 1427 | 1443
Not Completed | 66 | 70 | 83
Not completed — Adverse Event | 3 | 2 | 3
Not completed — Lost to Follow-up | 36 | 38 | 53
Not completed — As Per Sponsor Decision | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 27 | 30 | 25

BASELINE CHARACTERISTICS:
Groups:
- Inv_MMR_Min Group: Subjects received one dose of Inv_MMR, from a minimum potency lot (Inv_MMR_Min), co-administered with VV and HAV vaccines at Day 0. All US subjects were also co-administered PCV-13 vaccine. Approximately 6 weeks later, at Day 42, subjects were administered a dose from a separate lot of the Inv_MMR vaccine (Inv_MMR_Release), for the second dose. Inv_MMR and VV vaccines were administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- Inv_MMR_Med Group: Subjects received one dose of Inv_MMR, from a mid-range or medium potency lot (Inv_MMR_Med), co-administered with VV and HAV vaccines at Day 0. All US subjects were also co-administered PCV-13 vaccine. Approximately 6 weeks later, at Day 42, subjects were administered a dose from a separate lot of the Inv_MMR vaccine (Inv_MMR_Release), for the second dose. Inv_MMR and VV vaccines were administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- Com_MMR Group: Subjects received one dose of Com_MMR vaccine (Lot 1 or Lot 2), co-administered with VV and HAV vaccines at Day 0. All US subjects were also co-administered PCV-13 vaccine. Approximately 6 weeks later, at Day 42, subjects were administered a dose of Com_MMR vaccine (Lot 1 or Lot 2), for the second dose. Com_MMR and VV vaccines were administered subcutaneously in the triceps region of the left and right arm, respectively. HAV and PCV-13 vaccines were administered intramuscularly in the anterolateral region of the right and left thigh, respectively.
- Total: Total of all reporting groups
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group | Total
Number analyzed (Participants) | 1493 | 1497 | 1526 | 4516
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.6 (0.9) | 12.6 (0.9) | 12.6 (0.9) | 12.6 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 704 | 718 | 758 | 2180
  Male | 789 | 779 | 768 | 2336
Race/Ethnicity, Customized [Number; unit: Participants]
  African Heritage / African American | 45 | 53 | 46 | 144
  American Indian or Alaskan Native | 2 | 1 | 1 | 4
  Asian - Central/South Asian Heritage | 1 | 0 | 2 | 3
  Asian - East Asian Heritage | 3 | 0 | 1 | 4
  Asian - South East Asian Heritage | 362 | 366 | 367 | 1095
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  White - Arabic / North African Heritage | 8 | 8 | 8 | 24
  White - Caucasian / European Heritage | 1017 | 1022 | 1052 | 3091
  Other | 55 | 46 | 49 | 150

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value (by Enzyme-linked Immunosorbent Assay [ELISA])
Description: For measles virus, a seroresponse was defined as post-vaccination anti-measles virus antibody concentration equal or above [≥] 200 mIU/mL (ELISA) among subjects who were seronegative (antibody concentration less than [<] 150 mIU/mL) before dose 1. Criteria to demonstrate an acceptable immune response of Inv_MMR_Min/Inv_MMR_Med vaccine in terms of seroresponse rate for measles virus at Day 42: The lower limit of the two-sided 97.5% CI for the seroresponse rate of Inv_MMR_Min/Inv_MMR_Med was to be ≥ 90% for antibodies to measles virus.
Time Frame: At Day 42
Population: According-to-protocol (ATP) cohort for analysis of immunogenicity post dose 1: all eligible subjects with pre- & post-dose 1 serology results & were below assay cut-off for at least 1 vaccine antigen for MMR at pre-vaccination, did not meet elimination criteria up to Day 42 blood sample & complied with post-dose 1 blood sample schedule.
Measure: Number (97.5% Confidence Interval); unit: Percentage of subjects
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1361 | 1366 | 1378
Percentage of subjects
  Anti-measles ≥ 150 mIU/mL | 90.9 [89.0 to 92.6] | 94.3 [92.7 to 95.6] | 96.5 [95.2 to 97.5]
  Anti-measles ≥ 200 mIU/mL | 90.8 [88.9 to 92.5] | 94.2 [92.6 to 95.5] | 96.3 [95.0 to 97.3]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Min vaccine compared to Com_MMR vaccine in terms of seroresponse rate to measles virus at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% confidence interval (CI) on the group difference (Inv_MMR_Min minus Com_MMR) in seroresponse rate should be ≥ -5% for antibodies to measles virus when tested with ELISA; Difference in seroresponse rate = -5.48, 97.5% CI 2-sided [-7.65 to -3.43] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Med vaccine compared to Com_MMR vaccine in terms of seroresponse rate to measles virus at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% confidence interval (CI) on the group difference (Inv_MMR_Med minus Com_MMR) in seroresponse rate should be ≥ -5% for antibodies to measles virus when tested with ELISA; Difference in seroresponse rate = -2.08, 97.5% CI 2-sided [-3.96 to -0.27] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate

2. Primary Outcome: Percentage of Subjects With Anti-mumps Virus Antibody Concentration Equal to or Above the Cut-off-value (by ELISA)
Description: For mumps virus, a seroresponse was defined as post-vaccination anti-mumps virus antibody concentration ≥ 10 EU/mL (ELISA) among subjects who were seronegative (antibody concentration < 5 EU/mL) before dose 1. Criteria to demonstrate an acceptable immune response of Inv_MMR_Min/Inv_MMR_Med vaccine in terms of seroresponse rate for mumps virus at Day 42: The lower limit of the two-sided 97.5% CI for the seroresponse rate of Inv_MMR_Min/Inv_MMR_Med was to be ≥ 90% for antibodies to mumps virus.
Time Frame: At Day 42
Population: ATP cohort for analysis of immunogenicity post dose 1: all eligible subjects with pre- & post-dose 1 serology results & were below assay cut-off for at least 1 vaccine antigen for MMR at pre-vaccination, did not meet elimination criteria up to Day 42 blood sample & complied with post-dose 1 blood sample schedule.
Measure: Number (97.5% Confidence Interval); unit: Percentage of subjects
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1161 | 1131 | 1155
Percentage of subjects
  Anti-mumps ≥ 5 EU/mL | 99.1 [98.2 to 99.6] | 99.0 [98.1 to 99.6] | 99.2 [98.4 to 99.7]
  Anti-mumps ≥ 10 EU/mL | 97.4 [96.2 to 98.3] | 97.3 [96.0 to 98.2] | 97.8 [96.7 to 98.7]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Min vaccine compared to Com_MMR vaccine in terms of seroresponse rate to mumps virus at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group difference (Inv_MMR_Min minus Com_MMR) in seroresponse rate should be ≥ -5% for antibodies to mumps virus when tested with ELISA; Difference in seroresponse rate = -0.42, 97.5% CI 2-sided [-1.91 to 1.04] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Med vaccine compared to Com_MMR vaccine in terms of seroresponse rate to mumps virus at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group difference (Inv_MMR_Med minus Com_MMR) in seroresponse rate should be ≥ -5% for antibodies to mumps virus when tested with ELISA; Difference in seroresponse rate = -0.58, 97.5% CI 2-sided [-2.11 to 0.91] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate

3. Primary Outcome: Percentage of Subjects With Anti-mumps Virus Antibody Concentration Equal to or Above the Cut-off-value (by Plaque Reduction Neutralization Test [PRNT])
Description: For mumps virus as measured by PRNT, a seroresponse was defined as post-vaccination anti-mumps virus antibody concentration ≥ 4 End point Dilution 50% (ED50) (PRNT) among subjects who were seronegative (antibody concentration < 2.5 ED50) before dose 1.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1252 | 1265 | 1287
Percentage of subjects
  ≥ 2.5 ED50 | 79.1 [76.7 to 81.3] | 81.6 [79.3 to 83.7] | 87.5 [85.6 to 89.2]
  ≥ 4 ED50 | 71.2 [68.6 to 73.7] | 73.4 [70.8 to 75.8] | 80.6 [78.3 to 82.7]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group difference (Inv_MMR_Min minus Com_MMR) in seroresponse rate should be ≥ -10% for antibodies to mumps virus when tested with PRNT; Difference in seroresponse rate = -9.41, 97.5% CI 2-sided [-13.20 to -5.62] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; [analysis description as in outcome 2, analysis 2]; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group difference (Inv_MMR_Med minus Com_MMR) in seroresponse rate should be ≥ -10% for antibodies to mumps virus when tested with PRNT; Difference in seroresponse rate = -7.22, 97.5% CI 2-sided [-10.94 to -3.49] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate

4. Primary Outcome: Percentage of Subjects With Anti-rubella Virus Antibody Concentration Equal to or Above the Cut-off-value (by ELISA)
Description: For rubella virus, a seroresponse was defined as post-vaccination anti-rubella virus antibody concentration ≥ 10 IU/mL (ELISA) among subjects who were seronegative (antibody concentration < 4 IU/mL) before dose 1. Criteria to demonstrate an acceptable immune response of Inv_MMR_Min/Inv_MMR_Med vaccine in terms of seroresponse rate for rubella virus at Day 42: The lower limit of the two-sided 97.5% CI for the seroresponse rate of Inv_MMR_Min/Inv_MMR_Med was to be ≥ 90% for antibodies to mumps virus.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Number (97.5% Confidence Interval); unit: Percentage of subjects
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1359 | 1366 | 1376
Percentage of subjects
  ≥ 4 IU/mL | 99.3 [98.6 to 99.7] | 99.5 [98.9 to 99.8] | 99.5 [98.9 to 99.8]
  ≥ 10 IU/mL | 96.8 [95.5 to 97.7] | 97.3 [96.1 to 98.2] | 98.5 [97.6 to 99.1]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Min vaccine compared to Com_MMR vaccine in terms of seroresponse rate to rubella virus at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group difference (Inv_MMR_Min minus Com_MMR) in seroresponse rate should be ≥ -5% for antibodies to rubella virus when tested with ELISA; Difference in seroresponse rate = -1.71, 97.5% CI 2-sided [-3.11 to -0.42] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Med vaccine compared to Com_MMR vaccine in terms of seroresponse rate to rubella virus at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group difference (Inv_MMR_Med minus Com_MMR) in seroresponse rate should be ≥ -5% for antibodies to rubella virus when tested with ELISA; Difference in seroresponse rate = -1.18, 97.5% CI 2-sided [-2.50 to 0.05] — Asymptotic standardized 97.5% CI for the difference in seroresponse rate

5. Primary Outcome: Anti-measles Virus Antibody Concentrations (by ELISA)
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) in mIU/mL.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (97.5% Confidence Interval); unit: mIU/mL
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1361 | 1366 | 1378
mIU/mL | 2209.9 [2041.3 to 2392.4] | 2540.9 [2368.8 to 2725.5] | 2787.7 [2619.5 to 2966.7]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Min vaccine compared to COM_MMR vaccine in terms of GMCs for anti-measles antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Min over pooled Com_MMR) should to be ≥ 0.67 for antibodies to measles virus when tested with ELISA; ANOVA; 97.5% CI for GMC ratio was computed using ANOVA model on the log-transformed concentrations with vaccine group and the country as fixed effects; Adjusted GMC ratio = 0.79, 97.5% CI 2-sided [0.72 to 0.88]
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Med vaccine compared to COM_MMR vaccine in terms of GMCs for anti-measles antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Med over pooled Com_MMR) should to be ≥ 0.67 for antibodies to measles virus when tested with ELISA; ANOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 0.91, 97.5% CI 2-sided [0.83 to 1.01]

6. Primary Outcome: Anti-mumps Virus Antibody Concentrations (by ELISA)
Description: Antibody concentrations were expressed as GMCs in EU/mL.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (97.5% Confidence Interval); unit: EU/mL
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1161 | 1131 | 1155
EU/mL | 58.7 [55.5 to 62.1] | 60.2 [56.8 to 63.7] | 71.6 [67.7 to 75.8]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Min vaccine compared to COM_MMR vaccine in terms of GMCs for anti-mumps antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Min over pooled Com_MMR) should to be ≥ 0.67 for antibodies to mumps virus when tested with ELISA; ANOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 0.82, 97.5% CI 2-sided [0.76 to 0.89]
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Med vaccine compared to COM_MMR vaccine in terms of GMCs for anti-mumps antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Med over pooled Com_MMR) should to be ≥ 0.67 for antibodies to mumps virus when tested with ELISA; ANOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 0.84, 97.5% CI 2-sided [0.78 to 0.91]

7. Primary Outcome: Anti-mumps Virus Antibody Concentrations (by PRNT)
Description: Antibody concentrations were expressed as Geometric Mean Titers (GMTs).
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1252 | 1265 | 1287
Titers | 9.8 [9.0 to 10.6] | 10.7 [9.9 to 11.5] | 16.3 [15.1 to 17.7]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Min vaccine compared to COM_MMR vaccine in terms of GMCs for anti-mumps antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Min over pooled Com_MMR) should to be ≥ 0.67 for antibodies to mumps virus when tested with PRNT; ANOVA; 97.5% CI for GMC ratio was computed using ANOVA model on the log-transformed titers with vaccine group and the country as fixed effects; Adjusted GMT ratio = 0.60, 97.5% CI 2-sided [0.53 to 0.68]
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Med vaccine compared to COM_MMR vaccine in terms of GMCs for anti-mumps antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Med over pooled Com_MMR) should to be ≥ 0.67 for antibodies to mumps virus when tested with PRNT; ANOVA; [statistical method as in outcome 7, analysis 1]; Adjusted GMT ratio = 0.65, 97.5% CI 2-sided [0.57 to 0.74]

8. Primary Outcome: Anti-rubella Virus Antibody Concentrations (by ELISA)
Description: Antibody concentrations were expressed as GMCs in IU/mL.
Time Frame: At Day 42
Population: as for outcome 2
Measure: Geometric Mean (97.5% Confidence Interval); unit: IU/mL
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1359 | 1366 | 1376
IU/mL | 57.0 [54.1 to 60.0] | 56.9 [54.2 to 59.8] | 64.4 [61.4 to 67.5]
Statistical Analysis 1: Comparison: Inv_MMR_Min Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Min vaccine compared to COM_MMR vaccine in terms of GMCs for anti-rubella antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Min over pooled Com_MMR) should to be ≥ 0.67 for antibodies to rubella virus when tested with ELISA; ANOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 0.89, 97.5% CI 2-sided [0.83 to 0.95]
Statistical Analysis 2: Comparison: Inv_MMR_Med Group vs Com_MMR Group; Non-inferiority of Inv_MMR_Med vaccine compared to COM_MMR vaccine in terms of GMCs for anti-rubella antibodies at Day 42; Test type: Non-Inferiority — The lower limit of the 2-sided 97.5% CI on the group ratio of GMCs (Inv_MMR_Med over pooled Com_MMR) should to be ≥ 0.67 for antibodies to rubella virus when tested with ELISA; ANOVA; [statistical method as in outcome 5, analysis 1]; Adjusted GMC ratio = 0.88, 97.5% CI 2-sided [0.83 to 0.95]

9. Secondary Outcome: Percentage of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value (by ELISA)
Description: For measles virus, a seroresponse was defined as post-vaccination anti-measles virus antibody concentration ≥ 200 mIU/mL (ELISA) among subjects who were seronegative (antibody concentration < 150 mIU/mL) before dose 1.
Time Frame: At Day 84
Population: ATP cohort for analysis of immunogenicity post dose 2: all eligible subjects from US sub-cohort who received 2 doses of Inv_MMR/Com_MMR vaccine, with pre- & post-dose 2 serology results for at least 1 vaccine antigen for MMR, did not meet elimination criteria up to Day 84 blood sample & complied with post-dose 2 blood sample schedule.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 245 | 258 | 257
Percentage of subjects
  ≥ 150 mIU/mL | 99.6 [97.7 to 100] | 98.8 [96.6 to 99.8] | 98.8 [96.6 to 99.8]
  ≥ 200 mIU/mL | 99.6 [97.7 to 100] | 98.4 [96.1 to 99.6] | 98.4 [96.1 to 99.6]

10. Secondary Outcome: Percentage of Subjects With Anti-mumps Virus Antibody Concentration Equal to or Above the Cut-off-value (by ELISA)
Description: For mumps virus, a seroresponse was defined as post-vaccination anti-mumps virus antibody concentration ≥ 10 EU/mL (ELISA) among subjects who were seronegative (antibody concentration < 5 EU/mL) before dose 1.
Time Frame: At Day 84
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 216 | 199 | 212
Percentage of subjects
  ≥ 5 EU/mL | 99.1 [96.7 to 99.9] | 100 [98.2 to 100] | 99.1 [96.6 to 99.9]
  ≥ 10 EU/mL | 99.1 [96.7 to 99.9] | 100 [98.2 to 100] | 98.6 [95.9 to 99.7]

11. Secondary Outcome: Percentage of Subjects With Anti-rubella Virus Antibody Concentration Equal to or Above the Cut-off-value (by ELISA)
Description: For rubella virus, a seroresponse was defined as post-vaccination anti-rubella virus antibody concentration ≥ 10 IU/mL (ELISA) among subjects who were seronegative (antibody concentration < 4 IU/mL) before dose 1.
Time Frame: At Day 84
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 245 | 259 | 255
Percentage of subjects
  ≥ 4 IU/mL | 100 [98.5 to 100] | 100 [98.6 to 100] | 100 [98.6 to 100]
  ≥ 10 IU/mL | 99.6 [97.7 to 100] | 99.6 [97.9 to 100] | 99.6 [97.8 to 100]

12. Secondary Outcome: Anti-measles Virus Antibody Concentrations (by ELISA)
Description: Antibody concentrations were expressed as GMCs in mIU/mL.
Time Frame: At Day 84
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 245 | 258 | 257
mIU/mL | 4803.5 [4290.4 to 5378.0] | 4557.7 [4061.5 to 5114.4] | 4453.9 [3951.9 to 5019.8]

13. Secondary Outcome: Anti-mumps Virus Antibody Concentrations (by ELISA)
Description: Antibody concentrations were expressed as GMCs in EU/mL.
Time Frame: At Day 84
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 216 | 199 | 212
EU/mL | 88.9 [80.4 to 98.3] | 94.1 [85.3 to 103.8] | 86.4 [77.4 to 96.5]

14. Secondary Outcome: Anti-rubella Virus Antibody Concentrations (by ELISA)
Description: Antibody concentrations were expressed as GMCs in IU/mL.
Time Frame: At Day 84
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 245 | 259 | 255
IU/mL | 112.7 [104.1 to 122.0] | 110.7 [102.9 to 119.1] | 110.9 [101.8 to 120.8]

15. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs) Post Dose 1
Description: Assessed solicited local AEs were pain, redness and swelling. Any = Occurrence of the AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Total Vaccinated cohort (TVC) included all vaccinated subjects with at least one vaccine administration of either Inv_MMR lots or Com_MMR lots documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1453 | 1464 | 1482
Participants
  Any pain | 261 | 262 | 301
  Any redness | 232 | 256 | 286
  Any swelling | 89 | 97 | 122

16. Secondary Outcome: Number of Subjects With Any Solicited Local AEs Post Dose 2
Description: as for outcome 15
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: TVC included all vaccinated subjects with at least one vaccine administration of either Inv_MMR lots or Com_MMR lots documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1427 | 1440 | 1456
Participants
  Any pain | 170 | 183 | 196
  Any redness | 159 | 196 | 217
  Any swelling | 67 | 91 | 96

17. Secondary Outcome: Number of Subjects With Any Solicited General AEs Post Dose 1
Description: Assessed solicited general AEs were drowsiness, irritability/fussiness and loss of appetite. Any = Occurrence of the AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 15-day (Days 0-14) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1454 | 1466 | 1486
Participants
  Any drowsiness | 551 | 565 | 582
  Any irritability / fussiness | 749 | 792 | 788
  Any loss of appetite | 570 | 589 | 591

18. Secondary Outcome: Number of Subjects Reporting Any Fever Post Dose 1
Description: Any fever = Fever (axillary) ≥ 38°C.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1454 | 1466 | 1486
Participants | 582 | 617 | 618

19. Secondary Outcome: Number of Subjects Reporting Any Fever Post Dose 2
Description: Any fever = Fever (axillary) ≥ 38°C.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1426 | 1443 | 1455
Participants | 458 | 471 | 499

20. Secondary Outcome: Number of Subjects Reporting Any Rash Post Dose 1
Description: Assessed were any localized or generalized rash, rash with fever, varicella-like rash and measles/rubella-like rash. Any = Occurrence of the AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1454 | 1466 | 1486
Participants
  Any localized or generalized | 328 | 322 | 333
  Any with fever | 115 | 133 | 131
  Any varicella like | 57 | 53 | 45
  Any measles/rubella like | 53 | 61 | 68

21. Secondary Outcome: Number of Subjects Reporting Any Rash Post Dose 2
Description: as for outcome 20
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1426 | 1443 | 1455
Participants
  Any localized or generalized | 129 | 150 | 141
  Any with fever | 52 | 63 | 53
  Any varicella like | 0 | 0 | 1
  Any measles/rubella like | 22 | 14 | 14

22. Secondary Outcome: Number of Subjects Reporting Any MMR Specific Solicited General AEs Post Dose 1
Description: Assessed MMR specific solicited general AEs were any suspected signs of meningism including febrile convulsions and parotid/salivary gland swelling. Any = Occurrence of the AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1454 | 1466 | 1486
Participants
  Any parotid gland swelling | 3 | 2 | 3
  Any febrile convulsion | 3 | 4 | 3

23. Secondary Outcome: Number of Subjects Reporting Any MMR Specific Solicited General AEs Post Dose 2
Description: as for outcome 22
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1426 | 1443 | 1455
Participants
  Any parotid gland swelling | 1 | 2 | 0
  Any febrile convulsion | 2 | 6 | 4

24. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AES Post Dose 1
Description: Unsolicited AE was defined as any AE reported in reported in addition to those solicited during the clinical study and any solicited AE with onset outside the specified period of follow-up for solicited AEs. Any = Occurrence of the AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1493 | 1497 | 1526
Participants | 762 | 794 | 777

25. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AES Post Dose 2
Description: as for outcome 24
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1449 | 1464 | 1483
Participants | 667 | 703 | 690

26. Secondary Outcome: Number of Subjects Reporting Any AEs of Specific Interest
Description: AEs of specific interest included new onset chronic disease (NOCD) (e.g., autoimmune disorders, asthma, type I diabetes, vasculitis, celiac disease, conditions associated with sub-acute or chronic thrombocytopenia and allergies) and AEs prompting emergency room (ER) visits.
Time Frame: From Day 0 through the end of the study (Day 222)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1493 | 1497 | 1526
Participants
  Any NOCD | 35 | 39 | 33
  Any AE prompting ER visit | 348 | 361 | 347

27. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAEs assessed include any untoward medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity.
Time Frame: From Day 0 through the end of the study (Day 222)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
Number analyzed (Participants) | 1493 | 1497 | 1526
Participants | 91 | 102 | 92

ADVERSE EVENTS:
Time Frame: Solicited local & general AEs: During the 4-day (Days 0-3) and 15-day (Days 0-14) post-vaccination period, respectively; Unsolicited AEs: During the 43-day (Days 0-42) post-vaccination period; SAEs: From Day 0 through the end of the study (Day 222).
Arm/Group | Inv_MMR_Min Group | Inv_MMR_Med Group | Com_MMR Group
All-Cause Mortality (participants affected / at risk) | 1/1493 | 0/1497 | 1/1526
Serious Adverse Events (participants affected / at risk) | 91/1493 | 102/1497 | 92/1526
Other Adverse Events (participants affected / at risk) | 1299/1493 | 1311/1497 | 1330/1526
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inv_MMR_Min Group (N=1493) | Inv_MMR_Med Group (N=1497) | Com_MMR Group (N=1526)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Perianal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Teething (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Drowning (General disorders) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 6 (6) | 7 (7) | 2 (2)
Bronchitis (Infections and infestations) | 4 (5) | 10 (10) | 8 (8)
Bronchitis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Croup infectious (Infections and infestations) | 2 (2) | 3 (3) | 4 (4)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Encephalitis brain stem (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Exanthema subitum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 16 (16) | 19 (19) | 10 (10)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 6 (6) | 3 (3) | 7 (7)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
Herpangina (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Influenza (Infections and infestations) | 3 (3) | 2 (2) | 2 (2)
Laryngitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Laryngotracheitis obstructive (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nail bed infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 3 (4) | 3 (3) | 2 (2)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Otitis media viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otosalpingitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 2 (2) | 5 (5) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 14 (14) | 10 (10)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Pneumonia viral (Infections and infestations) | 2 (2) | 6 (7) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Accidental poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Child maltreatment syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 7 (7) | 6 (6)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 7 (8) | 13 (15) | 8 (8)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Henoch-schonlein purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inv_MMR_Min Group (N=1493) | Inv_MMR_Med Group (N=1497) | Com_MMR Group (N=1526)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (3) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Adenoiditis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Adenoviral conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 5 (5) | 4 (4)
Anal fissure (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Aphonia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 6 (6) | 7 (7) | 3 (3)
Application site erythema (General disorders) | 0 (0) | 1 (1) | 2 (2)
Application site hypersensitivity (General disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 24 (29) | 21 (23) | 12 (13)
Arthropod sting (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 5 (5) | 3 (3)
Balanoposthitis (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 1 (2)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (5) | 8 (9)
Bronchiolitis (Infections and infestations) | 18 (22) | 22 (22) | 21 (22)
Bronchitis (Infections and infestations) | 81 (92) | 96 (115) | 77 (95)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 2 (2)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bullous impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Burn infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
Campylobacter infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 6 (7) | 9 (9) | 7 (7)
Candida nappy rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 63 (67) | 79 (90) | 79 (87)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 2 (3) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (11) | 11 (13) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 8 (9) | 7 (8) | 9 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 59 (68) | 64 (74) | 75 (84)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Croup infectious (Infections and infestations) | 4 (4) | 11 (11) | 12 (13)
Crying (General disorders) | 4 (5) | 4 (4) | 5 (7)
Cryptosporidiosis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Decreased activity (General disorders) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 571 (575) | 593 (595) | 593 (593)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 9 (9) | 9 (10) | 17 (17)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 15 (16) | 14 (16) | 13 (15)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 12 (12) | 18 (19) | 21 (21)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 73 (83) | 71 (76) | 75 (80)
Disaccharide metabolism disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Ear canal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 19 (19) | 19 (20) | 12 (13)
Ear pain (Ear and labyrinth disorders) | 6 (6) | 7 (7) | 6 (6)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 16 (16) | 7 (7) | 7 (9)
Eczema impetiginous (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 19 (19) | 21 (23) | 19 (20)
Enterobiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 288 (394) | 331 (455) | 362 (505)
Erythema infectiosum (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Exanthema subitum (Infections and infestations) | 2 (2) | 5 (5) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Exposure to communicable disease (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 2 (2) | 3 (3)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Eye oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid bleeding (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (5) | 4 (4) | 7 (8)
Fatigue (General disorders) | 2 (2) | 2 (3) | 1 (1)
Feeding disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 1 (1)
Gastric ph decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Gastritis viral (Infections and infestations) | 3 (4) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 88 (93) | 95 (107) | 93 (100)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 7 (7) | 6 (6) | 9 (9)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Genital candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Genital labial adhesions (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 4 (5) | 4 (4) | 2 (2)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (3)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 10 (10) | 23 (23) | 10 (11)
Head injury (Injury, poisoning and procedural complications) | 8 (8) | 7 (7) | 7 (7)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 9 (9) | 8 (8) | 8 (8)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyposideraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 6 (6) | 7 (7) | 9 (9)
Inborn error of metabolism (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 7 (8) | 11 (13) | 10 (10)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 2 (3)
Injection site erythema (General disorders) | 11 (11) | 15 (15) | 9 (9)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 3 (3)
Injection site haemorrhage (General disorders) | 0 (0) | 3 (3) | 0 (0)
Injection site induration (General disorders) | 2 (2) | 4 (4) | 2 (2)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site mass (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 1 (1) | 1 (1)
Injection site papule (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 3 (3) | 5 (5) | 2 (2)
Injection site urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1)
Irritability (Psychiatric disorders) | 757 (781) | 795 (815) | 793 (815)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Keratosis follicular (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 6 (6) | 7 (7)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lactase deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Language disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 34 (35) | 34 (37) | 27 (30)
Lethargy (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0)
Lice infestation (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Lip disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 1 (1)
Lip ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 4 (5) | 5 (5)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 8 (8) | 5 (5) | 2 (2)
Macule (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 3 (3) | 2 (3) | 2 (4)
Malocclusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4) | 4 (4)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mycoplasma infection (Infections and infestations) | 5 (5) | 0 (0) | 1 (1)
Naevus flammeus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (12) | 10 (12)
Nasopharyngitis (Infections and infestations) | 148 (177) | 176 (210) | 134 (154)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 7 (7) | 1 (1) | 8 (8)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (6)
Otitis externa (Infections and infestations) | 5 (5) | 3 (3) | 3 (3)
Otitis media (Infections and infestations) | 95 (120) | 99 (117) | 116 (143)
Otitis media acute (Infections and infestations) | 46 (55) | 49 (60) | 57 (65)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 3 (4)
Pain (General disorders) | 334 (431) | 336 (445) | 378 (500)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Palatal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parasitic gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Penile adhesion (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 2 (2)
Penile erythema (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Perinatal brain damage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Perineal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 50 (61) | 53 (56) | 55 (57)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 14 (15) | 15 (16) | 17 (17)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 8 (8) | 9 (9)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Protein-losing gastroenteropathy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Pseudocroup (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Radial head dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Regurgitation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 4 (4) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 24 (25) | 24 (28) | 22 (30)
Respiratory tract infection viral (Infections and infestations) | 4 (5) | 9 (10) | 7 (11)
Restlessness (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 37 (53) | 49 (56) | 30 (33)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 32 (39) | 25 (33) | 39 (41)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Roseola (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 11 (12) | 10 (10) | 7 (7)
Sinusitis bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 5 (5)
Skin bacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin warm (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep phase rhythm disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 551 (552) | 567 (569) | 582 (582)
Spider naevus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 6 (6) | 3 (3)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 123 (156) | 152 (188) | 170 (218)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Tearfulness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 62 (86) | 71 (104) | 64 (82)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 4 (4)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tongue biting (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 34 (36) | 24 (27) | 34 (36)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 22 (31) | 17 (21) | 17 (22)
Tracheitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 350 (475) | 354 (473) | 365 (485)
Upper respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (3) | 4 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5) | 3 (3)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
Vaccination site erythema (General disorders) | 7 (7) | 6 (6) | 8 (8)
Vaccination site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site rash (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vaccination site swelling (General disorders) | 1 (1) | 1 (1) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Vessel puncture site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 45 (50) | 51 (57) | 57 (61)
Viral pharyngitis (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Viral tonsillitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (6) | 11 (12)
Vomiting (Gastrointestinal disorders) | 43 (55) | 42 (45) | 48 (51)
Vulvitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9) | 7 (7)
Wound (Injury, poisoning and procedural complications) | 4 (4) | 10 (10) | 5 (5)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.